CLINICAL TRIAL: NCT01272505
Title: Conventional SILS vs Harmonic Scalpel SILS
Acronym: SILS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSSILSVSCSILS
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2010-04

CONDITIONS: Gallbladde Stones

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- conventional SILC (Placebo Comparator): Conventional method of single incision laparoscopic cholecystectomy
  Interventions: Procedure: converntional SILC; Procedure: Harmonic scalpel Single incision laparoscopic cholecystectomy
- HS-SILC (Active Comparator)
  Interventions: Procedure: Harmonic scalpel Single incision laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: converntional SILC
  Arms: conventional SILC
Procedure: Harmonic scalpel Single incision laparoscopic cholecystectomy

SUMMARY:
Single incision laparoscopic cholecystectomy is gaining widespread acceptance. there are some obstacles making this procedure more complex than conventional laparoscopic cholecystectomy. The use of harmonic scalpel may aid in solving some of these issues that may allow simplification of the technique. The investigators will compare the ordinary method of single incision laparoscopic cholecystectomy versus harmonic scalpel single incision laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic gallbladder stones

Exclusion Criteria:

* acute cholecystitis cbd stones contraindications for laparoscopy

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 137 (Estimated)

PRIMARY OUTCOMES:
operative time

SECONDARY OUTCOMES:
complications

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura Gastroenterology Surgical Center, Al Mansurah, Dakahlia Governorate, Egypt